CLINICAL TRIAL: NCT02285231
Title: Anti-hyperglycemic Effect of Short-term Arginyl-fructose Supplementation in Subjects With Pre-diabetes and Newly Diagnosed Type 2 Diabetes: Randomized, Double-blinded, Placebo-controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, National Research Laboratory for Clinical Nutrigenetics/Nutrigenomics, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201406-BR-171-04
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Pre-diabetes
Keywords: Anti-hyperglycemic effect
MeSH Terms: conditions — Glucose Intolerance | interventions — fructosyl arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEST (Experimental): Arginyl-fructose Supplementation
  Interventions: Dietary Supplement: Arginyl-fructose
- Placebo (Experimental): Placebo Supplementation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Arginyl-fructose
  Arms: TEST
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
In this double-blind, placebo-controlled study, subjects with prediabetes and type 2 diabetes were randomly assigned to the placebo control group or the test (Arginyl-fructose: AF) group. We determined fasting serum levels of glucose, hemoglobin A1c (HbA1c), insulin, and free fatty acids (FFAs), were measured by 2-h oral glucose tolerance tests (OGTTs) at baseline and after the 6-week intervention.

ELIGIBILITY:
Inclusion Criteria:

- All subjects are with prediabetes (IFG or IGT) or newly diagnosed type 2 DM (T2DM) no taking medicine. IFG was defined as fasting glucose between 100 and 125 mg/dL and IGT was defined as 2-h OGTTs glucose levels 140-199 mg/dL. Newly diagnosed type 2 diabetes was defined as fasting glucose ≥126 mg/dL or 2-h OGTTs level ≥ 200 mg/dL.

Exclusion Criteria:

- Exclusion criteria included 1) glucose lowering medications or insulin injections; 2) abnormal liver or renal function; 3) chronic stomach and intestines disease; 4) chronic alcoholism; 5) pregnancy or intending to become pregnant during time of study. 6) complications; 7) an occupation that could be dangerous if hypoglycemia should occur.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
2-h oral glucose tolerance tests (OGTTs | 6 week

REFERENCES:
- [Derived] Park SE, Kim OH, Kwak JH, Lee KH, Kwon YI, Chung KH, Lee JH. Antihyperglycemic effect of short-term arginyl-fructose supplementation in subjects with prediabetes and newly diagnosed type 2 diabetes: randomized, double-blinded, placebo-controlled trial. Trials. 2015 Nov 14;16:521. doi: 10.1186/s13063-015-1036-z. PMID 26578409